CLINICAL TRIAL: NCT02222493
Title: A Phase 3 Randomized, Double-blind Study Assessing The Efficacy And Safety Of Pf-06438179 And Infliximab In Combination With Methotrexate In Subjects With Moderately To Severely Active Rheumatoid Arthritis Who Have Had An Inadequate Response To Methotrexate
Brief Title: A Study of PF-06438179 (Infliximab-Pfizer) and Infliximab in Combination With Methotrexate in Subjects With Active Rheumatoid Arthritis (REFLECTIONS B537-02).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B5371002; REFLECTIONS B537-02 (Other: Alias ID); 2013-004148-49 (EudraCT Number)
Record Dates: First submitted 2014-08-19; First posted 2014-08-21 (Estimated); Results first posted 2017-09-11 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Phase 3; infliximab; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GP1111; Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PF-06438179 (Experimental)
  Interventions: Biological: PF-06438179
- Infliximab (Active Comparator)
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: PF-06438179 — PF-06438179 will be administered by intravenous infusion at an initial dose of 3 mg/kg at 0, 2 and 6 weeks, then every 8 weeks.
  Other Names: Infliximab-Pfizer
  Arms: PF-06438179
Biological: Infliximab — Infliximab will be administered by intravenous infusion at an initial dose of 3 mg/kg at 0, 2 and 6 weeks, then every 8 weeks.
  Other Names: Infliximab-EU, Remicade
  Arms: Infliximab

SUMMARY:
The study will assess the efficacy and safety of PF-06438179 and infliximab in combination with methotrexate in subjects with active rheumatoid arthritis who have had an inadequate response to methotrexate.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of rheumatoid arthritis based on 2010 ACR/EULAR criteria for at least 4 months.

At least 6 tender (of 68 assessed) and 6 swollen (of 66 assessed) joints at screening and baseline.

HS-CRP equal or greater than 10 mg/L.

Must have received methotrexate for at least 12 weeks and be on a stable dose for at least 4 weeks.

Exclusion Criteria:

Evidence of untreated or inadequately treated latent or active TB.

Evidence or history of moderate or severe heart failure (NYHA Class III/IV)

Infection requiring hospitalization or parenteral antimicrobial therapy judged clinically significant by the investigator within 6 months prior to first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2014-08-26 (Actual); Primary Completion 2016-06-29 (Actual); Study Completion 2017-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (184):
- United States (43):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Clinical and Translational Research Center of Alabama, PC, Tuscaloosa, Alabama
  - Sun Valley Arthritis Center, Ltd., Peoria, Arizona
  - Arizona Arthritis & Rheumatology Associates, P.C., Phoenix, Arizona
  - St. Jude Hospital Yorba Linda DBA St. Joseph Heritage Healthcare, Fullerton, California
  - Arthritis & Osteoporosis Medical Center, La Palma, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - Desert Valley Medical Group, Victorville, California
  - Javed Rheumatology Associates, Inc, Newark, Delaware
  - Arthritis and Rheumatic Disease Specialties, Aventura, Florida
  - International Medical Research, Daytona Beach, Florida
  - Daytona Beach, Florida
  - San Marcus Research Clinic, Inc., Miami, Florida
  - Advance Medical Research Services Corporation, Miami, Florida
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - Alastair C. Kennedy, MD, Vero Beach, Florida
  - Indian River Primary Care, Vero Beach, Florida
  - Harbin Clinic, Rome, Georgia
  - Advanced Clinical Research, Meridian, Idaho
  - Methodist Medical Center of IL, Peoria, Illinois
  - Physician's Clinic of Iowa, P.C., Cedar Rapids, Iowa
  - Gilbert-Graves Clinic, Bowling Green, Kentucky
  - Graves-Gilbert Clinic Bowling Green, Bowling Green, Kentucky
  - Ochsner Clinic Baton Rouge, Baton Rouge, Louisiana
  - Arthritis and Diabetes Clinic, Inc., Monroe, Louisiana
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Western Michigan University Homer Stryker MD School of Medicine Center for Clinical Research, Battle Creek, Michigan
  - Arthritis, Rheumatic & Back Disease Associates, Voorhees Township, New Jersey
  - Trinity Health Center-Medical Arts, Minot, North Dakota
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading, LLC, Wyomissing, Pennsylvania
  - Low Country Rheumatology, PA, Charleston, South Carolina
  - Regional Health Clinical Research, Rapid City, South Dakota
  - Regional Medical Clinic, Rapid City, South Dakota
  - West Tennessee Research Institute, Jackson, Tennessee
  - Ramesh C Gupta, MD, Memphis, Tennessee
  - Austin Regional Clinic, Austin, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Accurate Clinical Research, Inc., Houston, Texas
  - Accurate Clinical Research, Nassau Bay, Texas
  - Pharmacy Services, Sentara Leigh Hospital, Norfolk, Virginia
  - Sentara Medical Group, Clinical Research, Norfolk, Virginia
  - The Seattle Arthritis Clinic, Seattle, Washington
- Australia (6):
  - Gold Coast Private Hospital Pty Ltd, Southport, Queensland
  - HPS Pharmacies, Southport, Queensland
  - Paradise Arthritis and Rheumatology Pty Ltd, Southport, Queensland
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - CliniPath Pathology, Osborne Park, Western Australia
  - R.K. Will Pty Ltd, Victoria Park, Western Australia
- Bosnia and Herzegovina (4):
  - Clinical Center University of Sarajevo, Sarajevo, Kanton Sarajevo
  - General Hospital "Prim.dr.Abdulah Nakas", Sarajevo, Kanton Sarajevo
  - University Clinical Center Tuzla, Tuzla, Tuzlanski Kanton
  - University Hospital Clinical Center Banja Luka, Banja Luka
- Brazil (2):
  - CETI - Centro de Estudos em Terapias Inovadoras, Curitiba, Paraná
  - Hospital Israelita Albert Einstein, São Paulo
- Bulgaria (3):
  - Multiprofile Hospital for Active Treatment Trimontium OOD, Plovdiv
  - University Multiprofile Hospital for Active Treatment (UMHAT) "Kaspela" EOOD, Plovdiv
  - University Multiprofile Hospital for Active Treatment (UMHAT) "Sv. Ivan Rilski" EAD, Sofia
- Clinical Research and Arthritis Center, Windsor, Ontario, Canada
- Czechia (8):
  - CCBR Czech Brno, s.r.o., Brno
  - Lekarna Lancier, s.r.o., Brno
  - BENU Lekarna, Pardubice
  - CCBR-SYNARC a.s., Pardubice
  - CCBR Czech Prague, s.r.o., Prague
  - Lekarna U Robina, s.r.o., Prague
  - Lekarna Hradebni s.r.o., Uherské Hradiště
  - MEDICAL PLUS, s.r.o., Uherské Hradiště
- Georgia (6):
  - LTD Tbilisi Central Hospital, Tbilisi
  - LTD Unimedi Kakheti, Tbilisi
  - Tbilisi Heart and Vascular Clinic LTD, Tbilisi
  - LTD MediClubGeorgia, Tbilisi
  - LTD Adapti, Tbilisi
  - LTD Medulla" Chemotherapy and Immunotherapy Clinic, Tbilisi
- Germany (5):
  - Schlosspark-Klinik, Berlin
  - Klinikum der Universität München, München
  - Elisabeth-Klinik gGmbH, Olsberg
  - Knappschaftsklinikum Saar GmbH, Püttlingen
  - Rheumazentrum Ratingen, Ratingen
- Guatemala (4):
  - Clínica Médica Especializada en Medicina Interna y Reumatología, Guatemala City
  - Clínica Médica especializada en Medicina Interna, Guatemala City
  - Centro de Nutricion y Rehabilitacion Cardiorespiratoria, S.A. (NUCARE), Guatemala City
  - Therapeutic Research Institute and Lab S.A, Guatemala City
- Hungary (2):
  - DRC Gyógyszervizsgáló Központ Kft., Balatonfüred
  - Qualiclinic Kft., Budapest
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Organization, Hadassah Medical Center, Ein-Karem, Jerusalem
  - Meir Medical Center, Kfar Saba
- Japan (23):
  - Anjo Kosei Hospital, Anjo-shi, Aichi-ken
  - Aso Iizuka Hospital, Iiduka, Fukuoka
  - Inoue Hospital, Takasaki, Gunma
  - Mazda Hospital, Aki-gun, Hiroshima
  - Sapporo City General Hospital, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Matsubara Mayflower Hospital, Katoh, Hyōgo
  - National Hospital Organization Sagamihara National Hospital, Sagamihara, Kanagawa
  - Yokohama Minami Kyosai Hospital, Yokohama, Kanagawa
  - National Hospital Organization Nagasaki Medical Center, Ōmura, Nagasaki
  - Sasebo Chuo Hospital, Sasebo, Nagasaki
  - Kurashiki Sweet Hospital, Kurashiki, Okayama-ken
  - Yuaikai Tomishiro Central Hospital, Tomigusuku, Okinawa
  - Saitama Medical Center, Kawagoe-shi, Saitama
  - Hirose Clinic, Tokorozawa-shi, Saitama
  - National Hospital Organization Shizuoka Medical Center, Sunto-gun, Shizuoka
  - St. Luke's International Hospital, Chuo-ku, Tokyo
  - Toho University Ohashi Medical Center, Meguro-ku, Tokyo
  - Showa University Hospital, Shinagawa-ku, Tokyo
  - National Hospital Organization Chiba-East Hospital, Chiba
  - Kondo clinic for rheumatism and orthopaedics, Fukuoka
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Kumamoto Orthopaedic Hospital, Kumamoto
- Jordan (2):
  - Jordan Hospital, Amman
  - King Abdullah University Hospital, Irbid
- LSMUL Kauno klinikos, Kaunas, Lithuania
- Mexico (3):
  - Centro de Alta Especialidad en Reumatología e Investigación del Potosí, S.C., San Luis de Potosí, SAN LUIS de Potosi
  - Unidad de Investigaciones Reumatológicas A.C - Hospital Central "Dr. Ignacio Morones Prieto", Zona Universitaria, SAN LUIS de Potosi
  - Unidad Reumatologica Las Americas S.C.P, Mérida, Yucatán
- Morocco (3):
  - El Ayachi Hospital, Salé
  - Groupe Radiologique de Salé, Salé
  - Laboratoire les Arcades d'Analyses Médicales, Salé
- Peru (7):
  - Hospital María Auxiliadora - Centro de Investigaciones Medicas, San Juan de Miraflores, Lima region
  - Instituto de Ginecología y Reproducción & Cirugía Mínimamente Invasiva, Santiago de Surco, Lima region
  - Centro de diagnóstico por imágenes, Radiología General y Especial, Arequipa
  - Unidad de Investigación en Medicina Interna y Enfermedades Críticas, Arequipa
  - Centro de Investigación Reumatología CAA, Lima
  - Clinica Medica Cayetano Heredia, Lima
  - Servicio de Inmunología y Reumatología, Lima
- Philippines (6):
  - Mary Mediatrix Medical Center, Lipa City, Batangas
  - Southern Philippines Medical Center, Davao City, Davao DEL SUR
  - Makati Medical Center, Makati City, National Capital Region
  - Medical Center Manila, Manila
  - Philippine General Hospital, Manila
  - St. Luke's Medical Center, Quezon
- Poland (5):
  - Szpital Uniwersytecki nr 2 im. dr. Jana Biziela w Bydgoszczy, Bydgoszcz
  - Szpital Specjalistyczny im. J. Dietla Malopolskie Centrum Reumatologii Immunologii i Rehabilitacji, Krakow
  - NZOZ Lecznica MAK-MED. S.C., Nadarzyn
  - Twoja Przychodnia - Centrum Medyczne Nowa Sol, Nowa Sól
  - MTZ Clinical Research Sp. z o.o., Warsaw
- Romania (3):
  - Spitalul Clinic Judetean de Urgenta Galati "Sf. Apostol Andrei", Galati
  - Spitalul Clinic de Recuperare Iasi, Iași
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Târgu Mureş
- Russia (14):
  - GBUZ "Republican hospital n.a. V.A.Baranov", Petrozavodsk, Republic of Karelia
  - GAUZ of Kemerovo Region "Regional clinical hospital for war veterans", Kemerovo
  - KGBUZ "Krasnoyarsk Interdistrict Clinical Hospital #20 n.a. I.S.Berzon", Krasnoyarsk
  - Krasnoyarsk State Medical University n.a.Prof.V.F.Voyno-Yasenetsky, Krasnoyarsk
  - GMU " Kursk regional clinical hospital" of the Committee of Healthcare of the Kursk region, Kursk
  - GBUZ of city of Moscow, Moscow
  - GBOU VPO "Ryazan State medical university n.a. academician I.P.Pavlov", Ryazan
  - GBOUVPO "Ryazan State Medical University n.a. Academician I.P.Pavlov", Ryazan
  - GBU of Ryazan region "Regional clinical cardiology dispanser", Ryazan
  - GBOU of Ryazan region "Regional clinical hospital", Ryazan
  - Spb GBUZ "Clinical rheumatology hospital # 25" City CDC prevention of osteoporosis, Saint Petersburg
  - GUZ "Regional clinical hospital", Saratov
  - GBUZ VO 'Regional clinical hospital", Vladimir
  - GBKUZ of Yaroslavl region "City hospital n. a. N.A. Semashko", Yaroslavl
- Serbia (3):
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Military Medical Academy, Belgrade
  - Institute for Treatment and Rehabilitation "Niska Banja", Niška Banja
- South Africa (5):
  - Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng
  - Jakaranda Hospital, Pretoria, Gauteng
  - Emmed Research, Pretoria, Gauteng
  - Arthritis Clinical Research Unit, Cape Town, Western Cape
  - Vincent Pallotti Hospital, Cape Town, Western Cape
- South Korea (6):
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Konkuk University Medical Center, Seoul
- Tunisia (2):
  - Mohamed Kassab Institute of orthopedics, Manouba
  - Rabta Hospital, Tunis
- Ukraine (12):
  - Derzhavna ustanova "Ukrainskyi derzhavnyi naukovo-doslidnyi instytut, Dnipropetrovsk
  - Oblasna klinichna likarnia, revmatolohichne viddilennia, Derzhavnyi vyshchyi navchalnyi zaklad, Ivano-Frankivsk
  - Komunalnyi zaklad okhorony zdorovia "Kharkivska miska klinichna likarnia #8", Kharkiv
  - Khmelnytska oblasna likarnia, Khmelnytskyi
  - Kyivska miska klinichna likarnia #6, Kyiv
  - Klinichnyi hospital Derzhavnoi prykordonnoi sluzhby Ukrainy, Lviv
  - Komunalnyi zaklad "Kryvorizka miska klinichna likarnia #2" Dnipropetrovskoi oblasnoi rady", M. Kryvyi Rih
  - Komunalnyi zaklad Sumskoi oblasnoi rady "Sumska oblasna klinichna likarnia", M. Sumy
  - Vinnytska oblasna klinichna likarnia im. M.I.Pyrohova, revmatolohichne, M. Vinnytsia
  - Komunalna ustanova "Odeska oblasna klinichna likarnia", Odesa
  - Bahatoprofilnyi medychnyi tsentr (Universytetska klinika #1), Odesa
  - Komunalna ustanova "Zaporizka oblasna klinichna likarnia" Zaporizkoi oblasnoi rady, Zaporizhzhia
- United Kingdom (2):
  - Wrightington Hospital, Wigan, Lancashire
  - Maidstone Hospital, Maidstone and Tunbridge wells NHS Trust, Maidstone

REFERENCES:
- [Derived] Kay J, Bock AE, Rehman M, Zhang W, Zhang M, Iikuni N, Alvarez DF. Use of multibiomarker disease activity scores in biosimilarity studies for the treatment of patients with rheumatoid arthritis. RMD Open. 2022 Sep;8(2):e002423. doi: 10.1136/rmdopen-2022-002423. PMID 36180101
- [Derived] Cohen SB, Radominski SC, Kameda H, Kivitz AJ, Tee M, Cronenberger C, Zhang M, Hackley S, Rehman MI, von Richter O, Alten R. Long-term Efficacy, Safety, and Immunogenicity of the Infliximab (IFX) Biosimilar, PF-06438179/GP1111, in Patients with Rheumatoid Arthritis After Switching from Reference IFX or Continuing Biosimilar Therapy: Week 54-78 Data From a Randomized, Double-Blind, Phase III Trial. BioDrugs. 2020 Apr;34(2):197-207. doi: 10.1007/s40259-019-00403-z. PMID 31939063
- [Derived] Palaparthy R, Rehman MI, von Richter O, Yin D. Population pharmacokinetics of PF-06438179/GP1111 (an infliximab biosimilar) and reference infliximab in patients with moderately to severely active rheumatoid arthritis. Expert Opin Biol Ther. 2019 Oct;19(10):1065-1074. doi: 10.1080/14712598.2019.1635583. Epub 2019 Jul 8. PMID 31284794
- [Derived] Alten R, Batko B, Hala T, Kameda H, Radominski SC, Tseluyko V, Babic G, Cronenberger C, Hackley S, Rehman M, von Richter O, Zhang M, Cohen S. Randomised, double-blind, phase III study comparing the infliximab biosimilar, PF-06438179/GP1111, with reference infliximab: efficacy, safety and immunogenicity from week 30 to week 54. RMD Open. 2019 Mar 28;5(1):e000876. doi: 10.1136/rmdopen-2018-000876. eCollection 2019. PMID 30997153
- [Derived] Cohen SB, Alten R, Kameda H, Hala T, Radominski SC, Rehman MI, Palaparthy R, Schumacher K, Schmitt S, Hua SY, Ianos C, Sewell KL. A randomized controlled trial comparing PF-06438179/GP1111 (an infliximab biosimilar) and infliximab reference product for treatment of moderate to severe active rheumatoid arthritis despite methotrexate therapy. Arthritis Res Ther. 2018 Jul 27;20(1):155. doi: 10.1186/s13075-018-1646-4. PMID 30053896
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5371002&StudyName=A%20Study%20of%20PF-06438179%20%28Infliximab-Pfizer%29%20and%20Infliximab%20in%20Combination%20with%20Methotrexate%20in%20Subjects%20with%20Active%20Rheumatoid%20Arthritis%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1603 participants were screened after signing an informed consent form, of whom 650 participants were randomized to receive study treatment. One (1) participant in the PF-06438179 arm was screened and randomized by 2 different study site personnel, and no data were collected for the participant's second randomization.
Groups:
- PF-06438179: Participants received intravenous infusions of PF-06438179 at 3 mg/kg on Weeks 0, 2, 6 followed by a maintenance dose every 8 weeks at Weeks 14 and 22 in Period 1 which ended with the completion of the Week 30 pre-dose assessments. For participants who failed to achieve a minimum clinical response or lost clinical response (after Week 14 assessments), dose was increased to 5 mg/kg per infusion every 8 weeks. Participants initially randomized to PF-06438179 continued to blindly receive PF-06438179 in Period 2. A second randomization was blindly performed prior to dosing at Week 30 (at the beginning of Period 2, when participants initially randomized to INX were re-randomized in a 1:1 ratio, with 50% of the participants switching to PF-06438179 and the other 50% of participants remaining on the INX arm. Period 3 started with dosing at Week 54 where all participants began open label treatment with PF-06438179.
- Infliximab-EU Remicade (INX): Participants received intravenous infusions of INX at 3 mg/kg on Weeks 0, 2, 6 followed by a maintenance dose every 8 weeks at Weeks 14 and 22 in Period 1 which ended with the completion of the Week 30 pre-dose assessments. For participants who failed to achieve a minimum clinical response or lost clinical response (after Week 14 assessments), dose was increased to 5 mg/kg per infusion every 8 weeks. Participants initially randomized to PF-06438179 continued to blindly receive PF-06438179 in Period 2. A second randomization was blindly performed prior to dosing at Week 30 (at the beginning of Period 2), when participants initially randomized to INX were re-randomized in a 1:1 ratio, with 50% of the participants switching to PF-06438179 and the other 50% of participants remaining on the INX arm. Period 3 started with dosing at Week 54 where all participants began open label treatment with PF-06438179.
Period: Period 1: First Dose-Week 30 (Pre-dose)
Arm/Group | PF-06438179 | Infliximab-EU Remicade (INX)
Started | 324 | 326
Received Treatment | 323 | 326
Completed | 280 | 286
Not Completed | 44 | 40
Not completed — Death | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 11 | 9
Not completed — Protocol Violation | 5 | 1
Not completed — Insufficient clinical response | 0 | 7
Not completed — Non-compliance with study treatment | 1 | 0
Not completed — Pregnancy | 2 | 0
Not completed — Adverse Event | 18 | 20
Not completed — Other | 4 | 0
Not completed — Randomized but not treated | 1 | 0
Period: Period 2: Week30 Dosing-Week54(Pre-dose)
Arm/Group | PF-06438179 | Infliximab-EU Remicade (INX)
Started | 423 | 143
Completed | 380 | 126
Not Completed | 43 | 17
Not completed — Death | 1 | 0
Not completed — Adverse Event | 22 | 9
Not completed — Other | 3 | 0
Not completed — Non-compliance with study treatment | 1 | 0
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Insufficient clinical response | 9 | 3
Period: Period 3: Week 54 Dosing-Week 78 Visit
Arm/Group | PF-06438179 | Infliximab-EU Remicade (INX)
Started | 505 | 0
Completed | 474 | 0
Not Completed | 31 | 0
Not completed — Insufficient clinical response | 3 | 0
Not completed — Adverse Event | 14 | 0
Not completed — Other | 4 | 0
Not completed — Non-compliance with study treatment | 1 | 0
Not completed — Withdrawal by Subject | 9 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) Population was defined as all participants who were randomized to study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-06438179 | Infliximab-EU Remicade (INX) | Total
Number analyzed (Participants) | 324 | 326 | 650
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (13.3) | 52.8 (12.9) | 52.8 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 258 | 264 | 522
  Male | 66 | 62 | 128

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 14: Period 1
Description: ACR20 response: greater than or equal to (>=) 20 percent (%) improvement in tender joint count (TJC); >= 20% improvement in swollen joint count (SJC); and >= 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity (PGA); physician global assessment of disease activity; self-assessed disability (health assessment questionnaire-disability index [HAQ-DI]); and C-Reactive Protein (CRP).
Time Frame: Week 14
Population: The ITT Population was defined as all participants who were randomized to study treatment. The primary analyses for ACR20 at Week 14 were performed with the missing data imputed using a non-responder imputation method.
Measure: Number; unit: participants
Groups:
- Period 1: PF-06438179: Participants were scheduled to receive intravenous infusions of PF-06438179 at a dose of 3 mg/kg on Weeks 0, 2, 6 followed by a maintenance dose every 8 weeks at Weeks 14 and 22 in Period 1 which ended with the completion of the Week 30 pre-dose assessment. For participants who failed to achieve a minimum clinical response or lost clinical response (after Week 14 assessments), dose was increased to 5 mg/kg per infusion every 8 weeks.
- Period 1: Infliximab-EU Remicade (INX): Participants were scheduled to receive intravenous infusions of INX at a dose of 3 mg/kg on Weeks 0, 2, 6 followed by a maintenance dose every 8 weeks at Weeks 14 and 22 in Period 1 which ended with the completion of the Week 30 pre-dose assessment. For participants who failed to achieve a minimum clinical response or lost clinical response (after Week 14 assessments), dose was increased to 5 mg/kg per infusion every 8 weeks.
Arm/Group | Period 1: PF-06438179 | Period 1: Infliximab-EU Remicade (INX)
Number analyzed (Participants) | 324 | 326
participants | 198 | 207
Statistical Analysis 1: Comparison: Period 1: PF-06438179 vs Period 1: Infliximab-EU Remicade (INX); Score statistic method; Test type: Non-Inferiority or Equivalence — Equivalence test; Proportion Difference = -2.39, 95% CI 2-sided [-9.92 to 5.11]
Statistical Analysis 2: Comparison: Period 1: PF-06438179 vs Period 1: Infliximab-EU Remicade (INX); Score statistic method; Test type: Non-Inferiority or Equivalence — Equivalence test; Proportion Difference = -2.39, 90% CI 2-sided [-8.75 to 4.02]

2. Secondary Outcome: Number of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 2, 4, 6, 12, 22 and 30 (Pre-dose): Period 1
Description: ACR20 response: >=20% improvement in tender joint count; >=20% improvement in swollen joint count; and >=20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; HAQ-DI and CRP.
Time Frame: Week 2, 4, 6, 12, 22 and 30 (pre-dose)
Population: The ITT Population was defined as all participants who were randomized to study treatment.
Measure: Number; unit: participants
Arm/Group | Period 1: PF-06438179 | Period 1: Infliximab-EU Remicade (INX)
Number analyzed (Participants) | 324 | 326
participants
  Week 2 | 105 | 121
  Week 4 | 170 | 190
  Week 6 | 187 | 201
  Week 12 | 210 | 214
  week 22 | 205 | 213
  Week 30 (pre-dose) | 197 | 209

3. Secondary Outcome: Number of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 38, 46 and 54 (Pre-dose): Period 2
Description: as for outcome 2
Time Frame: Week 38, 46 and 54 (pre-dose)
Population: The ITT Population was defined as all participants who were randomized to study treatment.
Measure: Number; unit: participants
Groups:
- Period 2: PF-06438179/PF-06438179: Participants randomized to receive intravenous infusions of PF-06438179 in Period 1 were scheduled to receive PF-06438179 in Period 2 at a dose of 3 mg/kg or 5 mg/kg on Weeks 30, 38 and 46. Period 2 ended with the completion of the Week 54 pre-dose assessments.
- Period 2: INX/INX: Participants randomized to receive intravenous infusions of INX in Period 1 were scheduled to receive INX in Period 2 at a dose of 3 mg/kg or 5 mg/kg on Weeks 30, 38 and 46. Period 2 ended with the completion of the Week 54 pre-dose assessments.
- Period 2: INX/PF-06438179: Participants randomized to receive intravenous infusions of INX in Period 1 were scheduled to receive PF-06438179 in Period 2 at a dose of 3 mg/kg or 5 mg/kg on Weeks 30, 38 and 46. Period 2 ended with the completion of the Week 54 pre-dose assessments.
Arm/Group | Period 2: PF-06438179/PF-06438179 | Period 2: INX/INX | Period 2: INX/PF-06438179
Number analyzed (Participants) | 280 | 143 | 143
participants
  Week 38 | 206 | 101 | 110
  Week 46 | 199 | 98 | 99
  Week 54 (pre-dose) | 199 | 92 | 101

4. Secondary Outcome: Number of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 62, 70 and 78: Period 3
Description: as for outcome 2
Time Frame: Week 62, 70 and 78
Population: The ITT population included all participants enrolled and treated with at least 1 dose of study treatment in Period 3.
Measure: Number; unit: participants
Groups:
- Period 3: PF-06438179/PF-06438179/PF-06438179: Participants received intravenous infusions of PF-06438179 in Period 1 and Period 2. In Period 3 they were scheduled to receive PF-06438179 at a dose of 3 mg/kg or 5 mg/kg on Weeks 54, 62 and 70. Period 3 ended at Week 78.
- Period 3: INX/INX/PF-06438179: Participants received intravenous infusions of INX in Period 1 and Period 2. In Period 3 they were scheduled to receive PF-06438179 at a dose of 3 mg/kg or 5 mg/kg on Weeks 54, 62 and 70. Period 3 ended at Week 78.
- Period 3: INX/PF-06438179/PF-06438179: Participants received intravenous infusions of INX in Period 1 and PF-06438179 in Period 2. In Period 3 they were scheduled to receive PF-06438179 at a dose of 3 mg/kg or 5 mg/kg on Weeks 54, 62 and 70. Period 3 ended at Week 78.
Arm/Group | Period 3: PF-06438179/PF-06438179/PF-06438179 | Period 3: INX/INX/PF-06438179 | Period 3: INX/PF-06438179/PF-06438179
Number analyzed (Participants) | 253 | 126 | 126
participants
  Week 62 | 199 | 89 | 103
  Week 70 | 199 | 87 | 98
  Week 78 | 192 | 86 | 98

5. Secondary Outcome: Number of Participants With an American College of Rheumatology 50% (ACR50) and ACR 70% Response at Week 2, 4, 6, 12, 14, 22 and 30 (Pre-dose): Period 1
Description: ACR50 response: >=50% improvement in tender joint count, >=50% improvement in swollen joint count improvement and >=50% in at least 3 of 5 remaining ACR core measures: participant assessment of pain, participant global assessment of disease activity, physician global assessment of disease activity, HAQ-DI and CRP. ACR70 response: >=70% improvement in tender joint count, >=70% improvement in swollen joint count improvement and >=70% in at least 3 of 5 remaining ACR core measures: participant assessment of pain, participant global assessment of disease activity, physician global assessment of disease activity, HAQ-DI and CRP.
Time Frame: Week 2, 4, 6, 12, 14, 22 and 30 (pre-dose)
Population: The ITT Population was defined as all participants who were randomized to study treatment.
Measure: Number; unit: participants
Arm/Group | Period 1: PF-06438179 | Period 1: Infliximab-EU Remicade (INX)
Number analyzed (Participants) | 324 | 326
participants
  ACR50 (Week 2) | 24 | 24
  ACR50 (Week 4) | 72 | 59
  ACR50 (Week 6) | 88 | 80
  ACR50 (Week 12) | 95 | 101
  ACR50 (Week 14) | 116 | 108
  ACR50 (Week 22) | 126 | 116
  ACR50 (Week 30, pre-dose) | 125 | 132
  ACR70 (Week 2) | 6 | 6
  ACR70 (Week 4) | 22 | 13
  ACR70 (Week 6) | 33 | 16
  ACR70 (Week 12) | 46 | 40
  ACR70 (Week 14) | 56 | 33
  ACR70 (Week 22) | 56 | 45
  ACR70 (Week 30, pre-dose) | 67 | 58

6. Secondary Outcome: Number of Participants With an American College of Rheumatology 50% (ACR50) and ACR 70% Response at Week 38, 46 and 54 (Pre-dose): Period 2
Description: as for outcome 5
Time Frame: Week 38, 46 and 54 (pre-dose)
Population: The ITT Population was defined as all participants who were randomized to study treatment.
Measure: Number; unit: participants
Arm/Group | Period 2: PF-06438179/PF-06438179 | Period 2: INX/INX | Period 2: INX/PF-06438179
Number analyzed (Participants) | 280 | 143 | 143
participants
  ACR50 (Week 38) | 132 | 58 | 75
  ACR50 (Week 46) | 135 | 55 | 63
  ACR50 (Week 54, pre-dose) | 135 | 61 | 65
  ACR70 (Week 38) | 77 | 33 | 38
  ACR70 (Week 46) | 75 | 33 | 33
  ACR70 (Week 54, pre-dose) | 82 | 33 | 35

7. Secondary Outcome: Number of Participants With an American College of Rheumatology 50% (ACR50) and ACR 70% Response at Week 62, 70 and 78: Period 3
Description: as for outcome 5
Time Frame: Week 62, 70 and 78
Population: The ITT population included all participants enrolled and treated with at least 1 dose of study treatment in Period 3.
Measure: Number; unit: participants
Arm/Group | Period 3: PF-06438179/PF-06438179/PF-06438179 | Period 3: INX/INX/PF-06438179 | Period 3: INX/PF-06438179/PF-06438179
Number analyzed (Participants) | 253 | 126 | 126
participants
  ACR50 (Week 62) | 132 | 59 | 71
  ACR50 (Week 70) | 142 | 61 | 67
  ACR50 (Week 78) | 150 | 57 | 73
  ACR70 (Week 62) | 88 | 31 | 41
  ACR70 (Week 70) | 92 | 35 | 44
  ACR70 (Week 78) | 98 | 33 | 44

8. Secondary Outcome: Change From Baseline in Disease Activity Score-CRP (4 Variables) (DAS28-4 [CRP]) and HAQ-DI at Week 2, 4, 6, 12, 14, 22 and 30: Period 1
Description: DAS28 is measure of disease activity in participants. DAS28-4 (CRP): calculated from SJC, TJC, CRP(mg/L) and PGA (participant rated disease activity on visual analogue scale [VAS] from 0 to 100 mm; high score=worse health). Total score range of DAS28-4 (CRP): 0 to 9.4(0=no activity; 9.4=extreme disease activity), higher score=more disease activity. DAS28-4(CRP) less than (<)2.6=remission, <3.2=low disease activity, >=3.2-5.1=moderate disease activity and greater than (>) 5.1=high disease activity. HAQ-DI assess degree of difficulty a participant experienced (past week) in 8 domain of daily activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip and other activities. Each item scored on a 4-point scale ranging from 0 to 3(0=no difficulty; 3=extreme difficulty). Overall score: sum of domain scores/number of domains answered. Total possible score range (0=least difficulty; 3=extreme difficulty); high scores=more difficulty in performing daily living activities.
Time Frame: Baseline (Day 1), Week 2, 4, 6, 12, 14, 22 and 30
Population: The ITT Population was defined as all participants who were randomized to study treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 1: PF-06438179 | Period 1: Infliximab-EU Remicade (INX)
Number analyzed (Participants) | 324 | 326
units on a scale
  DAS28-CRP (Baseline): number analyzed (Participants) | 321 | 325
  DAS28-CRP (Baseline) | 5.950 (0.9577) | 5.983 (0.9210)
  DAS28-CRP (Change at Week 2): number analyzed (Participants) | 318 | 324
  DAS28-CRP (Change at Week 2) | -1.213 (0.9280) | -1.241 (0.8879)
  DAS28-CRP (Change at Week 4): number analyzed (Participants) | 312 | 315
  DAS28-CRP (Change at Week 4) | -1.596 (1.1259) | -1.605 (1.0881)
  DAS28-CRP (Change at Week 6): number analyzed (Participants) | 312 | 319
  DAS28-CRP (Change at Week 6) | -1.710 (1.1959) | -1.750 (1.0885)
  DAS28-CRP (Change at Week 12): number analyzed (Participants) | 310 | 316
  DAS28-CRP (Change at Week 12) | -1.898 (1.3516) | -1.885 (1.2142)
  DAS28-CRP (Change at Week 14): number analyzed (Participants) | 310 | 314
  DAS28-CRP (Change at Week 14) | -1.901 (1.4125) | -1.827 (1.3019)
  DAS28-CRP (Change at Week 22): number analyzed (Participants) | 301 | 307
  DAS28-CRP (Change at Week 22) | -2.005 (1.4236) | -2.002 (1.2972)
  DAS28-CRP (Change at Week 30): number analyzed (Participants) | 292 | 297
  DAS28-CRP (Change at Week 30) | -2.140 (1.4197) | -2.117 (1.2738)
  HAQ-DI (Baseline): number analyzed (Participants) | 321 | 325
  HAQ-DI (Baseline) | 1.623 (0.6485) | 1.586 (0.6490)
  HAQ-DI (Change at Week 2): number analyzed (Participants) | 320 | 324
  HAQ-DI (Change at Week 2) | -0.317 (0.4100) | -0.328 (0.4370)
  HAQ-DI (Change at Week 4): number analyzed (Participants) | 317 | 321
  HAQ-DI (Change at Week 4) | -0.472 (0.4728) | -0.477 (0.4861)
  HAQ-DI (Change at Week 6): number analyzed (Participants) | 314 | 320
  HAQ-DI (Change at Week 6) | -0.496 (0.5505) | -0.520 (0.5022)
  HAQ-DI (Change at Week 12): number analyzed (Participants) | 311 | 318
  HAQ-DI (Change at Week 12) | -0.535 (0.5795) | -0.524 (0.5857)
  HAQ-DI (Change at Week 14): number analyzed (Participants) | 311 | 316
  HAQ-DI (Change at Week 14) | -0.572 (0.5910) | -0.531 (0.5876)
  HAQ-DI (Change at Week 22): number analyzed (Participants) | 301 | 311
  HAQ-DI (Change at Week 22) | -0.588 (0.6061) | -0.569 (0.5958)
  HAQ-DI (Change at Week 30): number analyzed (Participants) | 294 | 298
  HAQ-DI (Change at Week 30) | -0.621 (0.6484) | -0.612 (0.6546)

9. Secondary Outcome: Change From Baseline in Disease Activity Score-CRP (4 Variables) (DAS28-4 [CRP]) and HAQ-DI at Week 38, 46 and 54: Period 2
Description: DAS28 is measure of disease activity in participants. DAS28-4 (CRP): calculated from SJC, TJC, CRP(mg/L) and PGA (participant rated disease activity on VAS from 0 to 100 millimeter [mm]; high score=worse health). Total score range of DAS28-4 (CRP): 0 to 9.4(0=no activity; 9.4=extreme disease activity), higher score=more disease activity. DAS28-4(CRP) <2.6=remission, <3.2=low disease activity, >=3.2-5.1=moderate disease activity and >5.1=high disease activity. HAQ-DI assess degree of difficulty a participant experienced (past week) in 8 domain of daily activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip and other activities. Each item scored on a 4-point scale ranging from 0 to 3(0=no difficulty; 3=extreme difficulty). Overall score: sum of domain scores/number of domains answered. Total possible score range (0=least difficulty; 3=extreme difficulty); high scores=more difficulty in performing daily living activities.
Time Frame: Baseline (Week 30 pre-dose), Week 38, 46 and 54
Population: The ITT Population was defined as all participants who were randomized to study treatment. Here, "Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 2: PF-06438179/PF-06438179 | Period 2: INX/INX | Period 2: INX/PF-06438179
Number analyzed (Participants) | 278 | 142 | 141
units on a scale
  DAS28-CRP (Baseline) | 3.765 (1.4629) | 3.819 (1.3624) | 3.781 (1.2547)
  DAS28-CRP (Change at Week 38): number analyzed (Participants) | 276 | 141 | 140
  DAS28-CRP (Change at Week 38) | -0.181 (0.9574) | 0.036 (0.8686) | -0.059 (0.8756)
  DAS28-CRP (Change at Week 46): number analyzed (Participants) | 266 | 138 | 133
  DAS28-CRP (Change at Week 46) | -0.228 (1.0453) | 0.048 (1.2584) | -0.017 (1.0692)
  DAS28-CRP (Change at Week 54): number analyzed (Participants) | 256 | 129 | 128
  DAS28-CRP (Change at Week 54) | -0.275 (1.1338) | -0.109 (1.1801) | -0.057 (1.2339)
  HAQ-DI (Change at Baseline) | 0.978 (0.7042) | 0.913 (0.6634) | 0.951 (0.6481)
  HAQ-DI (Change at Week 38): number analyzed (Participants) | 277 | 141 | 141
  HAQ-DI (Change at Week 38) | -0.019 (0.3328) | 0.019 (0.2889) | 0.007 (0.3688)
  HAQ-DI (Change at Week 46): number analyzed (Participants) | 269 | 138 | 133
  HAQ-DI (Change at Week 46) | -0.043 (0.3774) | 0.014 (0.3823) | 0.035 (0.4325)
  HAQ-DI (Change at Week 54): number analyzed (Participants) | 259 | 130 | 129
  HAQ-DI (Change at Week 54) | -0.026 (0.4407) | 0.017 (0.4399) | -0.044 (0.3881)

10. Secondary Outcome: Change From Baseline in Disease Activity Score-CRP (4 Variables) (DAS28-4 [CRP]) and HAQ-DI at Week 62, 70 and 78: Period 3
Description: DAS28 is measure of disease activity in participants. DAS28-4 (CRP): calculated from SJC, TJC, CRP(mg/L) and PGA (participant rated disease activity on VAS from 0 to 100 mm; high score=worse health). Total score range of DAS28-4 (CRP): 0 to 9.4(0=no activity; 9.4=extreme disease activity), higher score=more disease activity. DAS28-4(CRP) <2.6=remission, <3.2=low disease activity, >=3.2-5.1=moderate disease activity and >5.1=high disease activity. HAQ-DI assess degree of difficulty a participant experienced (past week) in 8 domain of daily activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip and other activities. Each item scored on a 4-point scale ranging from 0 to 3(0=no difficulty; 3=extreme difficulty). Overall score: sum of domain scores/number of domains answered. Total possible score range (0=least difficulty; 3=extreme difficulty); high scores=more difficulty in performing daily living activities.
Time Frame: Baseline (Week 54 pre-dose), Week 62, 70 and 78
Population: The ITT population included all participants enrolled and treated with at least 1 dose of study treatment in Period 3. Here, "Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 3: PF-06438179/PF-06438179/PF-06438179 | Period 3: INX/INX/PF-06438179 | Period 3: INX/PF-06438179/PF-06438179
Number analyzed (Participants) | 249 | 123 | 126
units on a scale
  DAS28-CRP (Baseline): number analyzed (Participants) | 249 | 123 | 124
  DAS28-CRP (Baseline) | 3.386 (1.3229) | 3.561 (1.3123) | 3.594 (1.2572)
  DAS28-CRP (Change at Week 62): number analyzed (Participants) | 249 | 123 | 124
  DAS28-CRP (Change at Week 62) | -0.072 (0.9150) | -0.004 (0.8190) | -0.154 (0.6840)
  DAS28-CRP (Change at Week 70): number analyzed (Participants) | 244 | 119 | 121
  DAS28-CRP (Change at Week 70) | -0.157 (0.9502) | -0.168 (0.8421) | -0.162 (0.7970)
  DAS28-CRP (Change at Week 78): number analyzed (Participants) | 239 | 114 | 118
  DAS28-CRP (Change at Week 78) | -0.236 (1.0361) | -0.269 (0.9759) | -0.215 (1.0584)
  HAQ-DI (Baseline) | 0.905 (0.7050) | 0.893 (0.6691) | 0.883 (0.6109)
  HAQ-DI (Change at Week 62): number analyzed (Participants) | 249 | 123 | 124
  HAQ-DI (Change at Week 62) | -0.024 (0.3126) | 0.021 (0.2989) | 0.008 (0.2942)
  HAQ-DI (Change at Week 70): number analyzed (Participants) | 244 | 119 | 122
  HAQ-DI (Change at Week 70) | -0.046 (0.3502) | -0.027 (0.2758) | 0.030 (0.2950)
  HAQ-DI (Change at Week 78): number analyzed (Participants) | 239 | 116 | 118
  HAQ-DI (Change at Week 78) | -0.079 (0.3869) | -0.022 (0.3521) | 0.001 (0.3800)

11. Secondary Outcome: Number of Participants Achieving American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) and Disease Activity Score (DAS <2.6) Remission: Period 1
Description: ACR/EULAR remission was considered if the scores on tender joint count, swollen joint count, hs-CRP (mg/dL), and patient's global assessment of arthritis (PGA) all were less than or equal to (=<) 1 or the score on the simplified disease activity index (SDAI) was =<3.3. SDAI was calculated as the sum of number of tender and swollen joint count (using 28 joints), PGA, physician global assessment, and CRP (mg/dL). PGA was assessed on a 10 mm VAS ranging from 0 (very well) to 10 (very poor), where higher scores indicate worse health condition. Physician global assessment was recorded on a 10 mm VAS ranging from 0 (very well) to 10 (very poor), where higher scores indicated more disease activity. DAS28 calculated from number of swollen joints and painful joints using the 28 joints count, CRP (mg/dL) and PGA using a 10 mm-VAS from 0 (very well) to 10 (very poor), where higher scores indicate worse health condition. DAS28 <3.2: low disease activity, DAS28 <2.6: remission.
Time Frame: Week 2, 4, 6, 12, 14, 22 and Week 30 (pre-dose)
Population: The ITT Population was defined as all participants who were randomized to study treatment.
Measure: Number; unit: participants
Arm/Group | Period 1: PF-06438179 | Period 1: Infliximab-EU Remicade (INX)
Number analyzed (Participants) | 324 | 326
participants
  ACR/EULAR remission (Week 2) | 2 | 3
  ACR/EULAR remission (Week 4) | 10 | 11
  ACR/EULAR remission (Week 6) | 12 | 10
  ACR/EULAR remission (Week 12) | 28 | 17
  ACR/EULAR remission (Week 14) | 27 | 22
  ACR/EULAR remission (Week 22) | 25 | 20
  ACR/EULAR remission (Week 30, pre-dose) | 30 | 23
  DAS remission (Week 2) | 9 | 17
  DAS remission (Week 4) | 28 | 32
  DAS remission (Week 6) | 40 | 35
  DAS remission (Week 12) | 52 | 44
  DAS remission (Week 14) | 53 | 43
  DAS remission (Week 22) | 58 | 50
  DAS remission (Week 30, pre-dose) | 62 | 54

12. Secondary Outcome: Number of Participants Achieving American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) and Disease Activity Score (DAS <2.6) Remission: Period 2
Description: ACR/EULAR remission was considered if the scores on tender joint count, swollen joint count, hs-CRP (mg/dL), and PGA all were =<1 or the score on the SDAI was =<3.3. SDAI was calculated as the sum of number of tender and swollen joint count (using 28 joints), PGA, physician global assessment, and CRP (mg/dL). PGA was assessed on a 10 mm VAS ranging from 0 (very well) to 10 (very poor), where higher scores indicate worse health condition. Physician global assessment was recorded on a 10 mm VAS ranging from 0 (very well) to 10 (very poor), where higher scores indicated more disease activity. DAS28 calculated from number of swollen joints and painful joints using the 28 joints count, CRP (mg/dL) and PGA using a 10 mm-VAS from 0 (very well) to 10 (very poor), where higher scores indicate worse health condition. DAS28 <3.2: low disease activity, DAS28 <2.6: remission.
Time Frame: Week 38, 46 and 54 (pre-dose)
Population: The ITT Population was defined as all participants who were randomized to study treatment.
Measure: Number; unit: participants
Arm/Group | Period 2: PF-06438179/PF-06438179 | Period 2: INX/INX | Period 2: INX/PF-06438179
Number analyzed (Participants) | 280 | 143 | 143
participants
  ACR/EULAR remission (Week 38) | 29 | 15 | 8
  ACR/EULAR remission (Week 46) | 39 | 15 | 7
  ACR/EULAR remission (Week 54, pre-dose) | 42 | 18 | 13
  DAS remission (Week 38) | 74 | 26 | 25
  DAS remission (Week 46) | 76 | 30 | 21
  DAS remission (Week 54, pre-dose) | 79 | 33 | 29

13. Secondary Outcome: Number of Participants Achieving American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) and Disease Activity Score (DAS <2.6) Remission: Period 3
Description: as for outcome 12
Time Frame: Week 62, 70 and 78
Population: The ITT population included all participants enrolled and treated with at least 1 dose of study treatment in Period 3.
Measure: Number; unit: participants
Arm/Group | Period 3: PF-06438179/PF-06438179/PF-06438179 | Period 3: INX/INX/PF-06438179 | Period 3: INX/PF-06438179/PF-06438179
Number analyzed (Participants) | 253 | 126 | 126
participants
  ACR/EULAR remission (Week 62) | 46 | 19 | 20
  ACR/EULAR remission (Week 70) | 50 | 18 | 19
  ACR/EULAR remission (Week 78) | 57 | 19 | 18
  DAS remission (Week 62) | 85 | 33 | 34
  DAS remission (Week 70) | 82 | 40 | 34
  DAS remission (Week 78) | 94 | 39 | 41

14. Secondary Outcome: Number of Participants With European League Against Rheumatism (EULAR) Response: Period 1
Description: EULAR response was based on DAS28 EULAR response criteria which was defined as good response = DAS28 change of >1.2 with DAS28 =<3.2; moderate response = DAS28 change of >0.6 to =<1.2 with DAS28 >3.2-5.1 and no-response = DAS28 change of =<0.6 with DAS28 >5.1.
Time Frame: Week 2, 4, 6, 12, 14, 22 and Week 30 (pre-dose)
Population: The ITT Population was defined as all participants who were randomized to study treatment.
Measure: Number; unit: participants
Arm/Group | Period 1: PF-06438179 | Period 1: Infliximab-EU Remicade (INX)
Number analyzed (Participants) | 324 | 326
participants
  Week 2 (good response): number analyzed (Participants) | 317 | 324
  Week 2 (good response) | 24 | 34
  Week 2 (moderate response): number analyzed (Participants) | 317 | 324
  Week 2 (moderate response) | 172 | 161
  Week 2 (no response): number analyzed (Participants) | 317 | 324
  Week 2 (no response) | 121 | 129
  Week 4 (good response): number analyzed (Participants) | 312 | 315
  Week 4 (good response) | 61 | 56
  Week 4 (moderate response): number analyzed (Participants) | 312 | 315
  Week 4 (moderate response) | 162 | 172
  Week 4 (no response): number analyzed (Participants) | 312 | 315
  Week 4 (no response) | 89 | 87
  Week 6 (good response): number analyzed (Participants) | 312 | 319
  Week 6 (good response) | 65 | 64
  Week 6 (moderate response): number analyzed (Participants) | 312 | 319
  Week 6 (moderate response) | 168 | 181
  Week 6 (no response): number analyzed (Participants) | 312 | 319
  Week 6 (no response) | 79 | 74
  Week 12 (good response): number analyzed (Participants) | 310 | 316
  Week 12 (good response) | 90 | 88
  Week 12 (moderate response): number analyzed (Participants) | 310 | 316
  Week 12 (moderate response) | 149 | 162
  Week 12 (no response): number analyzed (Participants) | 310 | 316
  Week 12 (no response) | 71 | 66
  Week 14 (good response): number analyzed (Participants) | 310 | 314
  Week 14 (good response) | 97 | 82
  Week 14 (moderate response): number analyzed (Participants) | 310 | 314
  Week 14 (moderate response) | 137 | 155
  Week 14 (no response): number analyzed (Participants) | 310 | 314
  Week 14 (no response) | 76 | 77
  Week 22 (good response): number analyzed (Participants) | 301 | 307
  Week 22 (good response) | 103 | 96
  Week 22 (moderate response): number analyzed (Participants) | 301 | 307
  Week 22 (moderate response) | 125 | 156
  Week 22 (no response): number analyzed (Participants) | 301 | 307
  Week 22 (no response) | 73 | 55
  Week 30 (good response): number analyzed (Participants) | 292 | 297
  Week 30 (good response) | 101 | 94
  Week 30 (moderate response): number analyzed (Participants) | 292 | 297
  Week 30 (moderate response) | 133 | 155
  Week 30 (no response): number analyzed (Participants) | 292 | 297
  Week 30 (no response) | 58 | 48

15. Secondary Outcome: Number of Participants With European League Against Rheumatism (EULAR) Response: Period 2
Description: as for outcome 14
Time Frame: Week 38, 46 and Week 54 (pre-dose)
Population: The ITT Population was defined as all participants who were randomized to study treatment.
Measure: Number; unit: participants
Arm/Group | Period 2: PF-06438179/PF-06438179 | Period 2: INX/INX | Period 2: INX/PF-06438179
Number analyzed (Participants) | 280 | 143 | 143
participants
  Week 38 (good response): number analyzed (Participants) | 276 | 141 | 140
  Week 38 (good response) | 110 | 51 | 49
  Week 38 (moderate response): number analyzed (Participants) | 276 | 141 | 140
  Week 38 (moderate response) | 132 | 62 | 66
  Week 38 (no response): number analyzed (Participants) | 276 | 141 | 140
  Week 38 (no response) | 34 | 28 | 25
  Week 46 (good response): number analyzed (Participants) | 266 | 138 | 133
  Week 46 (good response) | 107 | 46 | 49
  Week 46 (moderate response): number analyzed (Participants) | 266 | 138 | 133
  Week 46 (moderate response) | 126 | 64 | 67
  Week 46 (no response): number analyzed (Participants) | 266 | 138 | 133
  Week 46 (no response) | 33 | 28 | 17
  Week 54 (good response): number analyzed (Participants) | 256 | 129 | 128
  Week 54 (good response) | 118 | 53 | 50
  Week 54 (moderate response): number analyzed (Participants) | 256 | 129 | 128
  Week 54 (moderate response) | 109 | 56 | 62
  Week 54 (no response): number analyzed (Participants) | 256 | 129 | 128
  Week 54 (no response) | 29 | 20 | 16

16. Secondary Outcome: Number of Participants With European League Against Rheumatism (EULAR) Response: Period 3
Description: as for outcome 14
Time Frame: Week 62, 70 and Week 78
Population: The ITT population included all participants enrolled and treated with at least 1 dose of study treatment in Period 3.
Measure: Number; unit: participants
Arm/Group | Period 3: PF-06438179/PF-06438179/PF-06438179 | Period 3: INX/INX/PF-06438179 | Period 3: INX/PF-06438179/PF-06438179
Number analyzed (Participants) | 253 | 126 | 126
participants
  Week 62 (good response): number analyzed (Participants) | 249 | 123 | 124
  Week 62 (good response) | 122 | 50 | 57
  Week 62 (moderate response): number analyzed (Participants) | 249 | 123 | 124
  Week 62 (moderate response) | 102 | 56 | 54
  Week 62 (no response): number analyzed (Participants) | 249 | 123 | 124
  Week 62 (no response) | 25 | 17 | 13
  Week 70 (good response): number analyzed (Participants) | 244 | 119 | 121
  Week 70 (good response) | 127 | 56 | 52
  Week 70 (moderate response): number analyzed (Participants) | 244 | 119 | 121
  Week 70 (moderate response) | 92 | 48 | 54
  Week 70 (no response): number analyzed (Participants) | 244 | 119 | 121
  Week 70 (no response) | 25 | 15 | 15
  Week 78 (good response): number analyzed (Participants) | 239 | 114 | 118
  Week 78 (good response) | 133 | 58 | 57
  Week 78 (moderate response): number analyzed (Participants) | 239 | 114 | 118
  Week 78 (moderate response) | 84 | 45 | 53
  Week 78 (no response): number analyzed (Participants) | 239 | 114 | 118
  Week 78 (no response) | 22 | 11 | 8

17. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Treatment Related TEAEs: Period 1
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to Week 30 that were absent before treatment or that worsened relative to pre-treatment state. Treatment-related TEAE was any untoward medical occurrence attributed to study drug in a participant who received study drug. AEs included both serious and non-serious adverse events.
Time Frame: Baseline (Day 1) up to Week 30
Population: Safety population was defined as all participants who were randomized and received at least 1 dose of study treatment, analyzed by actual treatment received.
Measure: Number; unit: participants
Arm/Group | Period 1: PF-06438179 | Period 1: Infliximab-EU Remicade (INX)
Number analyzed (Participants) | 323 | 326
participants
  TEAEs | 185 | 176
  SAEs | 16 | 20
  Treatment related TEAEs | 81 | 75
  Treatment related SAEs | 4 | 4

18. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Treatment Related TEAEs: Period 2
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to Week 54 that were absent before treatment or that worsened relative to pre-treatment state. Treatment-related TEAE was any untoward medical occurrence attributed to study drug in a participant who received study drug. AEs included both serious and non-serious adverse events.
Time Frame: Baseline (Week 30 pre-dose) up to Week 54
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Period 2: PF-06438179/PF-06438179 | Period 2: INX/INX | Period 2: INX/PF-06438179
Number analyzed (Participants) | 280 | 143 | 143
participants
  TEAEs | 103 | 48 | 54
  SAEs | 13 | 11 | 4
  Treatment related TEAEs | 32 | 20 | 16
  Treatment related SAEs | 2 | 5 | 0

19. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Treatment Related TEAEs: Period 3
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to Week 78 that were absent before treatment or that worsened relative to pre-treatment state. Treatment-related TEAE was any untoward medical occurrence attributed to study drug in a participant who received study drug. AEs included both serious and non-serious adverse events.
Time Frame: Baseline (Week 54 pre-dose) up to Week 78
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Period 3: PF-06438179/PF-06438179/PF-06438179 | Period 3: INX/INX/PF-06438179 | Period 3: INX/PF-06438179/PF-06438179
Number analyzed (Participants) | 253 | 126 | 126
participants
  TEAEs | 73 | 38 | 37
  SAEs | 3 | 3 | 6
  Treatment related TEAEs | 22 | 10 | 8
  Treatment related SAEs | 0 | 1 | 3

20. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) of Grade 3 or Higher Severity: Period 1
Description: AEs were graded in accordance with National Cancer Institute (NCI) Common Terminology Criteria for AEs (CTCAE) Version 4.03 as Grades 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life threatening AEs and Grade 5= death related to AE. AEs of Grade 3 and higher severity are reported in this outcome measure.
Time Frame: Baseline (Day 1) up to Week 30
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Period 1: PF-06438179 | Period 1: Infliximab-EU Remicade (INX)
Number analyzed (Participants) | 323 | 326
participants
  TEAEs (Grade 3) | 34 | 34
  TEAEs (Grade 4) | 1 | 6
  TEAEs (Grade 5) | 2 | 1

21. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) of Grade 3 or Higher Severity: Period 2
Description: as for outcome 20
Time Frame: Baseline (Week 30 pre-dose) up to Week 54
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Period 2: PF-06438179/PF-06438179 | Period 2: INX/INX | Period 2: INX/PF-06438179
Number analyzed (Participants) | 280 | 143 | 143
participants
  TEAEs (Grade 3) | 17 | 10 | 6
  TEAEs (Grade 4) | 3 | 3 | 0
  TEAEs (Grade 5) | 1 | 0 | 0

22. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) of Grade 3 or Higher Severity: Period 3
Description: as for outcome 20
Time Frame: Baseline (Week 54 pre-dose) up to Week 78
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Period 3: PF-06438179/PF-06438179/PF-06438179 | Period 3: INX/INX/PF-06438179 | Period 3: INX/PF-06438179/PF-06438179
Number analyzed (Participants) | 253 | 126 | 126
participants
  TEAEs (Grade 3) | 4 | 3 | 7
  TEAEs (Grade 4) | 1 | 0 | 0
  TEAEs (Grade 5) | 0 | 0 | 0

23. Secondary Outcome: Number of Participants With Laboratory Abnormalities: Period 1
Description: Criteria for abnormality:hematology: hemoglobin, hematocrit, red blood cell count, lymphocytes, neutrophils: <0.8*lower limit of normal (LLN); platelets: >1.75*upper limit of normal (ULN); white blood cell count: <0.6*LLN; basophils, eosinophils, monocytes: >1.2*ULN. liver function: bilirubin: >1.5*ULN; aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase: >3.0*ULN; protein, albumin: <0.8*LLN></0>1.2*ULN; renal function:blood urea nitrogen,creatinine: >1.3*ULN; uric acid: >1.2*ULN; electrolytes: sodium, potassium, chloride, calcium, bicarbonate: <0.9*LLN,>1.1*ULN; urinalysis: pH<4.5, >8; glucose, protein, blood, ketones, urobilinogen, bilirubin, nitrite; Other(glucose: <0.6*LLN,>1.5*ULN). Participants with any laboratory abnormality in Period 1 were reported in this outcome measure.
Time Frame: Baseline (Day 1) up to Week 30
Population: Safety population was defined as all participants who are randomized and receive at least 1 dose of study treatment, analyzed by actual treatment received. Here, "Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Period 1: PF-06438179 | Period 1: Infliximab-EU Remicade (INX)
Number analyzed (Participants) | 321 | 325
participants | 245 | 237

24. Secondary Outcome: Number of Participants With Laboratory Abnormalities: Period 2
Description: Criteria for abnormality:hematology: hemoglobin, hematocrit, red blood cell count, lymphocytes, neutrophils: <0.8*lower limit of normal (LLN); platelets: >1.75*upper limit of normal (ULN); white blood cell count: <0.6*LLN; basophils, eosinophils, monocytes: >1.2*ULN. liver function: bilirubin: >1.5*ULN; aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase: >3.0*ULN; protein, albumin: <0.8*LLN></0>1.2*ULN; renal function:blood urea nitrogen,creatinine: >1.3*ULN; uric acid: >1.2*ULN; electrolytes: sodium, potassium, chloride, calcium, bicarbonate: <0.9*LLN,>1.1*ULN; urinalysis: pH<4.5, >8; glucose, protein, blood, ketones, urobilinogen, bilirubin, nitrite; Other(glucose: <0.6*LLN,>1.5*ULN). Participants with any laboratory abnormality in Period 2 were reported in this outcome measure.
Time Frame: Baseline (Week 30 pre-dose) up to Week 54
Population: as for outcome 23
Measure: Number; unit: participants
Arm/Group | Period 2: PF-06438179/PF-06438179 | Period 2: INX/INX | Period 2: INX/PF-06438179
Number analyzed (Participants) | 279 | 142 | 141
participants | 154 | 83 | 63

25. Secondary Outcome: Number of Participants With Laboratory Abnormalities: Period 3
Description: Criteria for abnormality:hematology: hemoglobin, hematocrit, red blood cell count, lymphocytes, neutrophils: <0.8*lower limit of normal (LLN); platelets: >1.75*upper limit of normal (ULN); white blood cell count: <0.6*LLN; basophils, eosinophils, monocytes: >1.2*ULN. liver function: bilirubin: >1.5*ULN; aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase: >3.0*ULN; protein, albumin: <0.8*LLN></0>1.2*ULN; renal function:blood urea nitrogen,creatinine: >1.3*ULN; uric acid: >1.2*ULN; electrolytes: sodium, potassium, chloride, calcium, bicarbonate: <0.9*LLN,>1.1*ULN; urinalysis: pH<4.5, >8; glucose, protein, blood, ketones, urobilinogen, bilirubin, nitrite; Other(glucose: <0.6*LLN,>1.5*ULN). Participants with any laboratory abnormality in Period 3 were reported in this outcome measure.
Time Frame: Baseline (Week 54 pre-dose) up to Week 78
Population: as for outcome 23
Measure: Number; unit: participants
Arm/Group | Period 3: PF-06438179/PF-06438179/PF-06438179 | Period 3: INX/INX/PF-06438179 | Period 3: INX/PF-06438179/PF-06438179
Number analyzed (Participants) | 250 | 123 | 126
participants | 127 | 72 | 61

26. Secondary Outcome: Change From Baseline in Tender Joint Count and Swollen Joint Count at Week 2, 4, 6, 12, 14, 22 and 30: Period 1
Description: Tender joint count was an assessment of 68 joints (upper body, upper extremity, and lower extremity). Each joint's response to pressure/motion was assessed as: Present or Absent. Swollen joint count was an assessment of 66 joints (upper body, upper extremity, and lower extremity). Each joint was assessed for swelling as: Present or Absent.
Time Frame: Baseline (Day 1), Week 2, 4, 6, 12, 14, 22 and Week 30
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Period 1: PF-06438179 | Period 1: Infliximab-EU Remicade (INX)
Number analyzed (Participants) | 321 | 325
joints
  Tender joint count (Baseline) | 24.7 (13.90) | 25.8 (12.89)
  Tender joint count (Change at Week 2): number analyzed (Participants) | 319 | 324
  Tender joint count (Change at Week 2) | -5.9 (8.78) | -7.5 (8.39)
  Tender joint count (Change at Week 4): number analyzed (Participants) | 317 | 321
  Tender joint count (Change at Week 4) | -9.5 (10.02) | -10.4 (9.41)
  Tender joint count (Change at Week 6): number analyzed (Participants) | 313 | 319
  Tender joint count (Change at Week 6) | -10.6 (11.17) | -12.1 (10.12)
  Tender joint count (Change at Week 12): number analyzed (Participants) | 311 | 318
  Tender joint count (Change at Week 12) | -12.1 (11.84) | -13.2 (11.51)
  Tender joint count (Change at Week 14): number analyzed (Participants) | 311 | 316
  Tender joint count (Change at Week 14) | -11.8 (12.50) | -13.0 (12.15)
  Tender joint count (Change at Week 22): number analyzed (Participants) | 301 | 311
  Tender joint count (Change at Week 22) | -13.2 (12.62) | -15.2 (12.93)
  Tender joint count (Change at Week 30): number analyzed (Participants) | 294 | 298
  Tender joint count (Change at Week 30) | -14.4 (13.19) | -15.6 (12.57)
  Swollen joint count (Baseline) | 16.1 (9.44) | 16.3 (8.70)
  Swollen joint count (Change at Week 2): number analyzed (Participants) | 319 | 324
  Swollen joint count (Change at Week 2) | -5.5 (6.89) | -5.7 (7.27)
  Swollen joint count (Change at Week 4): number analyzed (Participants) | 317 | 321
  Swollen joint count (Change at Week 4) | -7.8 (7.75) | -7.9 (7.39)
  Swollen joint count (Change at Week 6): number analyzed (Participants) | 313 | 319
  Swollen joint count (Change at Week 6) | -8.6 (7.99) | -9.0 (7.92)
  Swollen joint count (Change at Week 12): number analyzed (Participants) | 311 | 318
  Swollen joint count (Change at Week 12) | -9.6 (8.61) | -9.6 (8.39)
  Swollen joint count (Change at Week 14): number analyzed (Participants) | 311 | 316
  Swollen joint count (Change at Week 14) | -9.3 (8.87) | -9.6 (8.44)
  Swollen joint count (Change at Week 22): number analyzed (Participants) | 301 | 311
  Swollen joint count (Change at Week 22) | -10.5 (8.77) | -10.2 (7.94)
  Swollen joint count (Change at Week 30): number analyzed (Participants) | 294 | 298
  Swollen joint count (Change at Week 30) | -11.0 (9.33) | -10.7 (8.52)

27. Secondary Outcome: Change From Baseline in Tender Joint Count and Swollen Joint Count at Week 38, 46 and 54: Period 2
Description: as for outcome 26
Time Frame: Baseline (Week 30 pre-dose), Week 38, 46 and Week 54
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Period 2: PF-06438179/PF-06438179 | Period 2: INX/INX | Period 2: INX/PF-06438179
Number analyzed (Participants) | 278 | 142 | 141
joints
  Tender joint count (Baseline) | 10.2 (11.74) | 10.2 (11.96) | 9.1 (8.89)
  Tender joint count (Change at Week 38): number analyzed (Participants) | 277 | 141 | 141
  Tender joint count (Change at Week 38) | -1.3 (6.74) | -0.5 (8.86) | -1.0 (6.03)
  Tender joint count (Change at Week 46): number analyzed (Participants) | 269 | 138 | 133
  Tender joint count (Change at Week 46) | -1.6 (7.87) | -1.0 (9.32) | -0.8 (7.77)
  Tender joint count (Change at Week 54): number analyzed (Participants) | 260 | 130 | 129
  Tender joint count (Change at Week 54) | -1.7 (7.96) | -1.7 (10.23) | -0.5 (9.03)
  Swollen joint count (Baseline) | 4.9 (6.46) | 5.3 (6.57) | 4.6 (5.35)
  Swollen joint count (Change at Week 38): number analyzed (Participants) | 277 | 141 | 141
  Swollen joint count (Change at Week 38) | -0.8 (4.19) | -0.1 (4.90) | -0.3 (3.93)
  Swollen joint count (Change at Week 46): number analyzed (Participants) | 269 | 138 | 133
  Swollen joint count (Change at Week 46) | -1.2 (5.20) | 0.0 (5.54) | -0.5 (4.22)
  Swollen joint count (Change at Week 54): number analyzed (Participants) | 260 | 130 | 129
  Swollen joint count (Change at Week 54) | -1.3 (5.52) | -0.9 (7.02) | -0.7 (4.10)

28. Secondary Outcome: Change From Baseline in Tender Joint Count and Swollen Joint Count at Week 62, 70 and 78: Period 3
Description: as for outcome 26
Time Frame: Baseline (Week 54 pre-dose), Week 62, 70 and 78
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Period 3: PF-06438179/PF-06438179/PF-06438179 | Period 3: INX/INX/PF-06438179 | Period 3: INX/PF-06438179/PF-06438179
Number analyzed (Participants) | 249 | 123 | 126
joints
  Tender joint count (Baseline) | 7.5 (9.51) | 7.5 (9.21) | 7.4 (7.99)
  Tender joint count (Change at Week 62): number analyzed (Participants) | 249 | 123 | 124
  Tender joint count (Change at Week 62) | -0.7 (5.88) | 0.3 (5.21) | -0.8 (5.18)
  Tender joint count (Change at Week 70): number analyzed (Participants) | 244 | 119 | 122
  Tender joint count (Change at Week 70) | -1.4 (6.32) | -0.6 (5.14) | -1.0 (5.51)
  Tender joint count (Change at Week 78): number analyzed (Participants) | 239 | 116 | 118
  Tender joint count (Change at Week 78) | -1.7 (6.57) | -1.0 (5.82) | -1.4 (6.63)
  Swollen joint count (Baseline) | 3.4 (5.72) | 4.1 (5.16) | 3.5 (4.28)
  Swollen joint count (Change at Week 62): number analyzed (Participants) | 249 | 123 | 124
  Swollen joint count (Change at Week 62) | -0.3 (3.76) | 0.0 (4.41) | -0.3 (2.72)
  Swollen joint count (Change at Week 70): number analyzed (Participants) | 244 | 119 | 122
  Swollen joint count (Change at Week 70) | -0.7 (4.60) | -0.4 (4.12) | -0.5 (2.48)
  Swollen joint count (Change at Week 78): number analyzed (Participants) | 239 | 116 | 118
  Swollen joint count (Change at Week 78) | -0.9 (4.63) | -0.5 (4.00) | -0.2 (3.14)

29. Secondary Outcome: Change From Baseline in Patient's Assessment of Arthritis Pain (PAAP), Patient's Global Assessment of Arthritis (PGA) and Physician's Global Assessment of Arthritis (PGAA) at Week 2, 4, 6, 12, 14, 22, 30: Period 1
Description: PAAP: Participants assessed the severity of their arthritis pain by using a 100 mm VAS ranging from 0 (no pain) to 100 (most severe pain), which corresponded to the magnitude of their pain, where higher scores indicated more pain. PGA: Participants were asked the following question, "Considering all the ways your arthritis affects you, how are you feeling today?" and their response was recorded on a 100 mm VAS ranging from 0 (very well) to 100 (very poor), where higher scores indicated worse health condition. PGAA: Participants were assessed how their overall arthritis appears at the time of the visit. The evaluation was based on the participant's disease signs, functional capacity and physical examination, and was independent of the PAAP and PGA assessments. The physician's response was recorded using a 100 mm VAS ranging from 0 (very well) to 100 (very poor), where higher scores indicated more disease activity.
Time Frame: Baseline (Day 1), Week 2, 4, 6, 12, 14, 22 and 30
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 1: PF-06438179 | Period 1: Infliximab-EU Remicade (INX)
Number analyzed (Participants) | 321 | 325
units on a scale
  PAAP (Baseline) | 63.514 (20.5903) | 63.098 (21.5442)
  PAAP (Change at Week 2): number analyzed (Participants) | 320 | 324
  PAAP (Change at Week 2) | -15.724 (21.9589) | -15.360 (19.4328)
  PAAP (Change at Week 4): number analyzed (Participants) | 317 | 321
  PAAP (Change at Week 4) | -21.609 (22.3825) | -20.552 (21.2670)
  PAAP (Change at Week 6): number analyzed (Participants) | 314 | 320
  PAAP (Change at Week 6) | -23.917 (25.0213) | -22.797 (22.9133)
  PAAP (Change at Week 12): number analyzed (Participants) | 311 | 318
  PAAP (Change at Week 12) | -25.364 (25.6602) | -25.829 (24.8304)
  PAAP (Change at Week 14): number analyzed (Participants) | 311 | 316
  PAAP (Change at Week 14) | -26.131 (26.8712) | -25.077 (25.0536)
  PAAP (Change at week 22): number analyzed (Participants) | 301 | 311
  PAAP (Change at week 22) | -27.844 (27.0039) | -25.788 (25.3225)
  PAAP (Change at Week 30): number analyzed (Participants) | 294 | 298
  PAAP (Change at Week 30) | -29.150 (27.9802) | -28.853 (26.7252)
  PGA (Baseline) | 65.340 (20.7209) | 63.752 (22.9105)
  PGA (Change at Week 2): number analyzed (Participants) | 320 | 324
  PGA (Change at Week 2) | -17.262 (22.8767) | -16.504 (20.3188)
  PGA (Change at Week 4): number analyzed (Participants) | 317 | 321
  PGA (Change at Week 4) | -23.393 (23.3769) | -21.355 (23.6005)
  PGA (Change at Week 6): number analyzed (Participants) | 314 | 320
  PGA (Change at Week 6) | -25.536 (24.8041) | -23.314 (24.2005)
  PGA (Change at Week 12): number analyzed (Participants) | 311 | 317
  PGA (Change at Week 12) | -26.882 (25.3270) | -26.535 (26.3998)
  PGA (Change at Week 14): number analyzed (Participants) | 311 | 316
  PGA (Change at Week 14) | -27.583 (26.7955) | -25.323 (26.8562)
  PGA (Change at Week 22): number analyzed (Participants) | 301 | 310
  PGA (Change at Week 22) | -28.558 (27.5077) | -26.486 (26.7141)
  PGA (Change at Week 30): number analyzed (Participants) | 294 | 298
  PGA (Change at Week 30) | -29.186 (28.6488) | -28.814 (28.5929)
  PGAA (Baseline): number analyzed (Participants) | 319 | 325
  PGAA (Baseline) | 65.362 (16.2520) | 64.126 (16.7220)
  PGAA (Change at Week 2): number analyzed (Participants) | 318 | 324
  PGAA (Change at Week 2) | -21.913 (18.5574) | -20.143 (17.1407)
  PGAA (Change at Week 4): number analyzed (Participants) | 315 | 321
  PGAA (Change at Week 4) | -29.724 (19.2226) | -27.905 (17.9803)
  PGAA (Change at Week 6): number analyzed (Participants) | 312 | 320
  PGAA (Change at Week 6) | -33.319 (20.1143) | -30.958 (18.9303)
  PGAA (Change at Week 12): number analyzed (Participants) | 310 | 318
  PGAA (Change at Week 12) | -34.827 (19.8162) | -33.919 (19.7020)
  PGAA (Change at Week 14): number analyzed (Participants) | 310 | 316
  PGAA (Change at Week 14) | -35.870 (21.4707) | -34.175 (20.6526)
  PGAA (Change at Week 22): number analyzed (Participants) | 300 | 311
  PGAA (Change at Week 22) | -37.542 (20.8619) | -36.118 (20.6564)
  PGAA (Change at Week 30): number analyzed (Participants) | 293 | 298
  PGAA (Change at Week 30) | -39.842 (22.0276) | -36.666 (22.1598)

30. Secondary Outcome: Change From Baseline in Patient's Assessment of Arthritis Pain (PAAP), Patient's Global Assessment of Arthritis (PGA) and Physician's Global Assessment of Arthritis (PGAA) at Week 38, 46 and 54: Period 2
Description: as for outcome 29
Time Frame: Baseline (Week 30 pre-dose), Week 38, 46 and 54
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 2: PF-06438179/PF-06438179 | Period 2: INX/INX | Period 2: INX/PF-06438179
Number analyzed (Participants) | 278 | 142 | 141
units on a scale
  PAAP (Baseline) | 33.137 (24.2922) | 33.331 (22.2738) | 32.559 (22.2702)
  PAAP (Change at Week 38): number analyzed (Participants) | 277 | 141 | 141
  PAAP (Change at Week 38) | -0.014 (18.7502) | 1.440 (14.9902) | -0.705 (18.9147)
  PAAP (Change at Week 46): number analyzed (Participants) | 269 | 138 | 133
  PAAP (Change at Week 46) | -2.230 (20.0201) | 1.087 (21.5811) | 2.188 (20.7319)
  PAAP (Change at Week 54): number analyzed (Participants) | 259 | 130 | 129
  PAAP (Change at Week 54) | -1.416 (20.7823) | -0.492 (20.8000) | 1.365 (24.8362)
  PGA (Baseline) | 35.104 (24.8444) | 33.268 (22.2621) | 34.029 (22.7172)
  PGA (Change at Week 38): number analyzed (Participants) | 277 | 141 | 141
  PGA (Change at Week 38) | -1.628 (19.1471) | 1.582 (16.0776) | -1.086 (17.5787)
  PGA (Change at Week 46): number analyzed (Participants) | 269 | 138 | 133
  PGA (Change at Week 46) | -3.171 (20.3050) | 0.558 (20.6610) | 0.535 (21.3947)
  PGA (Change at Week 54): number analyzed (Participants) | 259 | 130 | 129
  PGA (Change at Week 54) | -2.929 (20.9396) | -0.538 (21.1331) | 0.776 (23.8743)
  PGAA (Baseline) | 25.124 (19.0943) | 27.294 (18.8148) | 26.091 (17.9503)
  PGAA (Change at Week 38): number analyzed (Participants) | 277 | 141 | 141
  PGAA (Change at Week 38) | -1.254 (12.4789) | 0.588 (16.5232) | -1.852 (15.4699)
  PGAA (Change at Week 46): number analyzed (Participants) | 269 | 138 | 133
  PGAA (Change at Week 46) | -2.470 (13.9135) | 0.625 (20.0163) | -0.700 (18.8038)
  PGAA (Change at Week 54): number analyzed (Participants) | 258 | 130 | 129
  PGAA (Change at Week 54) | -2.252 (17.0422) | -3.398 (20.0381) | -2.969 (20.1498)

31. Secondary Outcome: Change From Baseline in Patient's Assessment of Arthritis Pain (PAAP), Patient's Global Assessment of Arthritis (PGA) and Physician's Global Assessment of Arthritis (PGAA) at Week 62, 70 and 78: Period 3
Description: as for outcome 29
Time Frame: Baseline (Week 54 pre-dose), Week 62, 70 and 78
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 3: PF-06438179/PF-06438179/PF-06438179 | Period 3: INX/INX/PF-06438179 | Period 3: INX/PF-06438179/PF-06438179
Number analyzed (Participants) | 249 | 123 | 126
units on a scale
  PAAP (Baseline) | 30.395 (23.7412) | 31.659 (23.2900) | 31.225 (22.9366)
  PAAP (Change at Week 62): number analyzed (Participants) | 249 | 123 | 124
  PAAP (Change at Week 62) | -0.025 (15.8259) | 0.276 (12.2744) | -1.790 (16.6740)
  PAAP (Change at Week 70): number analyzed (Participants) | 244 | 118 | 122
  PAAP (Change at Week 70) | -2.948 (18.1105) | -0.297 (15.4108) | -0.970 (16.7170)
  PAAP (Change at Week 78): number analyzed (Participants) | 238 | 116 | 118
  PAAP (Change at Week 78) | -3.552 (18.8760) | -2.900 (18.0663) | -3.918 (20.9632)
  PGA (Baseline) | 30.841 (23.7807) | 31.130 (23.3603) | 32.710 (22.6365)
  PGA (Change at Week 62): number analyzed (Participants) | 249 | 123 | 124
  PGA (Change at Week 62) | 0.240 (16.2724) | 1.463 (13.6899) | -2.226 (15.3415)
  PGA (Change at Week 70): number analyzed (Participants) | 244 | 119 | 122
  PGA (Change at Week 70) | -1.764 (18.7038) | 0.101 (14.4260) | -2.093 (16.2677)
  PGA (Change at Week 78): number analyzed (Participants) | 239 | 115 | 118
  PGA (Change at Week 78) | -2.880 (19.6643) | -2.339 (17.0453) | -3.758 (19.5447)
  PGAA (Baseline) | 21.305 (17.6278) | 21.780 (17.3354) | 20.705 (16.9587)
  PGAA (Change at Week 62): number analyzed (Participants) | 249 | 123 | 124
  PGAA (Change at Week 62) | -0.381 (13.6810) | 2.659 (14.6314) | -0.499 (12.9483)
  PGAA (Change at Week 70): number analyzed (Participants) | 244 | 119 | 122
  PGAA (Change at Week 70) | -3.217 (14.1581) | -1.160 (12.7665) | -0.810 (15.0274)
  PGAA (Change at Week 78): number analyzed (Participants) | 239 | 116 | 118
  PGAA (Change at Week 78) | -2.217 (15.3894) | 0.681 (15.0989) | -0.159 (17.2024)

32. Secondary Outcome: Change From Baseline in High Sensitivity C-Reactive Protein (Hs-CRP) Concentration at Week 2, 4, 6, 12, 14, 22 and 30: Period 1
Time Frame: Baseline (Day 1), Week 2, 4, 6, 12, 14, 22 and 30
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milligram/litres
Arm/Group | Period 1: PF-06438179 | Period 1: Infliximab-EU Remicade (INX)
Number analyzed (Participants) | 321 | 325
milligram/litres
  Baseline | 25.916 (24.3118) | 25.366 (28.4866)
  Change at Week 2: number analyzed (Participants) | 318 | 324
  Change at Week 2 | -17.183 (20.8107) | -16.140 (24.2442)
  Change at Week 4: number analyzed (Participants) | 312 | 315
  Change at Week 4 | -15.555 (19.5227) | -13.407 (33.9136)
  Change at Week 6: number analyzed (Participants) | 313 | 320
  Change at Week 6 | -14.078 (20.4984) | -13.247 (27.7801)
  Change at Week 12: number analyzed (Participants) | 311 | 317
  Change at Week 12 | -12.502 (23.9435) | -12.525 (27.8736)
  Change at Week 14: number analyzed (Participants) | 310 | 314
  Change at Week 14 | -12.613 (23.2548) | -12.392 (29.3267)
  Change at Week 22: number analyzed (Participants) | 301 | 308
  Change at Week 22 | -11.195 (24.5225) | -11.422 (31.0610)
  Change at Week 30: number analyzed (Participants) | 292 | 297
  Change at Week 30 | -12.165 (25.6612) | -12.390 (30.0352)

33. Secondary Outcome: Change From Baseline in High Sensitivity C-Reactive Protein (Hs-CRP) Concentration at Week 38, 46 and 54: Period 2
Time Frame: Baseline (Week 30 pre-dose), Week 38, 46 and 54
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milligrams/litres
Arm/Group | Period 2: PF-06438179/PF-06438179 | Period 2: INX/INX | Period 2: INX/PF-06438179
Number analyzed (Participants) | 278 | 142 | 141
milligrams/litres
  Baseline | 12.970 (19.1927) | 14.427 (21.1595) | 10.847 (14.8018)
  Change at Week 38: number analyzed (Participants) | 276 | 141 | 140
  Change at Week 38 | 0.496 (18.7859) | 1.805 (19.5138) | 0.093 (14.8441)
  Change at Week 46: number analyzed (Participants) | 266 | 138 | 133
  Change at Week 46 | 1.210 (16.1727) | 3.996 (24.4986) | 0.798 (15.7687)
  Change at Week 54: number analyzed (Participants) | 256 | 129 | 128
  Change at Week 54 | 0.639 (21.1226) | 2.988 (24.5492) | 1.264 (13.6788)

34. Secondary Outcome: Change From Baseline in High Sensitivity C-Reactive Protein (Hs-CRP) Concentration at Week 62, 70 and 78: Period 3
Time Frame: Baseline (Week 54 pre-dose), Week 62, 70 and 78
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: milligrams/litres
Arm/Group | Period 3: PF-06438179/PF-06438179/PF-06438179 | Period 3: INX/INX/PF-06438179 | Period 3: INX/PF-06438179/PF-06438179
Number analyzed (Participants) | 249 | 123 | 126
milligrams/litres
  Baseline | 13.112 (21.3781) | 16.096 (24.1595) | 11.985 (13.8159)
  Change at Week 62: number analyzed (Participants) | 249 | 123 | 124
  Change at Week 62 | -0.635 (19.9660) | -3.648 (21.6177) | -0.541 (9.3198)
  Change at Week 70: number analyzed (Participants) | 244 | 119 | 121
  Change at Week 70 | -0.320 (23.1234) | -4.199 (22.3368) | -0.339 (11.7095)
  Change at Week 78: number analyzed (Participants) | 239 | 115 | 118
  Change at Week 78 | -1.660 (19.6340) | -3.565 (23.9800) | 0.811 (14.7061)

35. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADA) and Neutralizing Antibodies (Nab) Status: Period 1
Description: ADA positive results was defined as ADA titer level >=1.30 and NAb positive was defined as NAb titer level >=0.70.
Time Frame: Baseline (Day 1) up to Week 30
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Period 1: PF-06438179 | Period 1: Infliximab-EU Remicade (INX)
Number analyzed (Participants) | 323 | 326
participants
  ADA | 157 | 167
  NAb: number analyzed (Participants) | 157 | 167
  NAb | 124 | 143

36. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADA) and Neutralizing Antibodies (Nab) Status: Period 2
Description: ADA positive results was defined as ADA titer level >=1.30 and NAb positive was defined as NAb titer level >=0.70.
Time Frame: Baseline (Week 30 pre-dose) up to Week 54
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Period 2: PF-06438179/PF-06438179 | Period 2: INX/INX | Period 2: INX/PF-06438179
Number analyzed (Participants) | 280 | 143 | 143
participants
  ADA | 146 | 86 | 83
  NAb: number analyzed (Participants) | 146 | 86 | 83
  NAb | 118 | 73 | 65

37. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADA) and Neutralizing Antibodies (Nab) Status: Period 3
Description: ADA positive results was defined as ADA titer level >=1.30 and NAb positive was defined as NAb titer level >=0.70.
Time Frame: Baseline (Week 54 pre-dose) up to Week 78
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Period 3: PF-06438179/PF-06438179/PF-06438179 | Period 3: INX/INX/PF-06438179 | Period 3: INX/PF-06438179/PF-06438179
Number analyzed (Participants) | 253 | 126 | 126
participants
  ADA | 119 | 66 | 72
  NAb: number analyzed (Participants) | 119 | 66 | 72
  NAb | 105 | 58 | 60

38. Secondary Outcome: Serum Concentration Versus Time Summary: Period 1
Time Frame: Pre dose on Day 1, 15, 43, 99, 155 and 211; 2 hours post dose on Day 1 and 99; and 336 hours post dose on Day 29
Population: Pharmacokinetic population: all treated participants from per protocol (PP) population, who had at least 1 post-dose drug concentration measurement during Period 1. PP population: all participants who were randomized and received the study treatment as planned up to Week 14, with no major protocol deviations.
Measure: Median (Standard Deviation); unit: nanograms/milliliters
Groups:
- Period 1: Infliximab-EU Remicade (INX): Participants were scheduled to receive intravenous infusions INX at a dose of 3 mg/kg on Weeks 0, 2, 6 followed by a maintenance dose every 8 weeks at Weeks 14 and 22 in Period 1 which ended with the completion of the Week 30 pre-dose assessment. For participants who failed to achieve a minimum clinical response or lost clinical response (after Week 14 assessments), dose was increased to 5 mg/kg per infusion every 8 weeks.
Arm/Group | Period 1: PF-06438179 | Period 1: Infliximab-EU Remicade (INX)
Number analyzed (Participants) | 323 | 326
nanograms/milliliters
  Day 1 (0 hours): number analyzed (Participants) | 322 | 323
  Day 1 (0 hours) | 1635 (11163) | 656.2 (6583.8)
  Day 1 (2 hours): number analyzed (Participants) | 319 | 322
  Day 1 (2 hours) | 65310 (24920) | 62220 (22129)
  Day 15 (0 hours): number analyzed (Participants) | 316 | 323
  Day 15 (0 hours) | 17350 (8391.4) | 16690 (8002.7)
  Day 29 (336 hours): number analyzed (Participants) | 308 | 314
  Day 29 (336 hours) | 23640 (12357) | 21570 (10986)
  Day 43 (0 hours): number analyzed (Participants) | 308 | 315
  Day 43 (0 hours) | 11440 (10101) | 10100 (7721.7)
  Day 99 (0 hours): number analyzed (Participants) | 302 | 310
  Day 99 (0 hours) | 3547 (9559.2) | 2559 (6360.3)
  Day 99 (2 hours): number analyzed (Participants) | 297 | 299
  Day 99 (2 hours) | 76030 (39407) | 73350 (41410)
  Day 155 (0 hours): number analyzed (Participants) | 295 | 303
  Day 155 (0 hours) | 2051 (3440.9) | 1566 (2321.4)
  Day 211 (0 hours): number analyzed (Participants) | 281 | 290
  Day 211 (0 hours) | 1781 (2765.2) | 2112 (11703)

39. Secondary Outcome: Serum Concentration Versus Time Summary: Period 2
Time Frame: Pre dose on Day 211, 267, 379 and 547
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: nanograms/milliliters
Arm/Group | Period 2: PF-06438179/PF-06438179 | Period 2: INX/INX | Period 2: INX/PF-06438179
Number analyzed (Participants) | 280 | 143 | 143
nanograms/milliliters
  Day 211 (0 hours): number analyzed (Participants) | 278 | 143 | 142
  Day 211 (0 hours) | 1801 (2773.4) | 1083 (1763.6) | 1819 (2393.5)
  Day 267 (0 hours): number analyzed (Participants) | 272 | 136 | 133
  Day 267 (0 hours) | 1855 (2871.7) | 1208 (1926.5) | 1620 (2413.7)
  Day 379 (0 hours): number analyzed (Participants) | 248 | 125 | 125
  Day 379 (0 hours) | 2075 (4054.6) | 1823 (6110.8) | 1734 (2725.2)
  Day 547 (0 hours): number analyzed (Participants) | 16 | 14 | 11
  Day 547 (0 hours) | 499.6 (1373.0) | 212.7 (405.18) | 3305 (8429.5)

40. Secondary Outcome: Serum Concentration Versus Time Summary: Period 3
Time Frame: Pre dose on Day 379, 435 and 547
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: nanograms/milliliters
Arm/Group | Period 3: PF-06438179/PF-06438179/PF-06438179 | Period 3: INX/INX/PF-06438179 | Period 3: INX/PF-06438179/PF-06438179
Number analyzed (Participants) | 253 | 126 | 126
nanograms/milliliters
  Day 379 (0 hours): number analyzed (Participants) | 250 | 125 | 125
  Day 379 (0 hours) | 2078 (4044.0) | 1823 (6110.8) | 1734 (2725.2)
  Day 435 (0 hours): number analyzed (Participants) | 243 | 118 | 123
  Day 435 (0 hours) | 1913 (2838.0) | 1388 (2387.4) | 1572 (2543.4)
  Day 547: number analyzed (Participants) | 243 | 121 | 119
  Day 547 | 1707 (2512.9) | 1663 (5305.7) | 1482 (2441.6)

ADVERSE EVENTS:
Time Frame: Period 1: Baseline (Day 1) up to Week 30, Period 2: Baseline (Week 30 pre-dose) up to Week 54, Period 3: Baseline (Week 54 pre-dose) up to Week 78
Description: Safety population was defined as all participants who are randomized and receive at least 1 dose of study treatment, analyzed by actual treatment received. The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non serious in another participant, or 1 participant may have experienced both a serious and non serious event during the study.
Arm/Group | Period 1: PF-06438179 | Period 1: Infliximab-EU Remicade (INX) | Period 2: PF-06438179/PF-06438179 | Period 2: INX/INX | Period 2: INX/PF-06438179 | Period 3: PF-06438179/PF-06438179/PF-06438179 | Period 3: INX/INX/PF-06438179 | Period 3: INX/PF-06438179/PF-06438179
Serious Adverse Events (participants affected / at risk) | 16/323 | 20/326 | 13/280 | 11/143 | 4/143 | 3/253 | 3/126 | 6/126
Other Adverse Events (participants affected / at risk) | 38/323 | 35/326 | 8/280 | 11/143 | 6/143 | 0/253 | 0/126 | 0/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: PF-06438179 (N=323) | Period 1: Infliximab-EU Remicade (INX) (N=326) | Period 2: PF-06438179/PF-06438179 (N=280) | Period 2: INX/INX (N=143) | Period 2: INX/PF-06438179 (N=143) | Period 3: PF-06438179/PF-06438179/PF-06438179 (N=253) | Period 3: INX/INX/PF-06438179 (N=126) | Period 3: INX/PF-06438179/PF-06438179 (N=126)
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Keratitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multi-organ disorder (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Purulent synovitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Venous stenosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood disorder (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ocular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Genital prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bone abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: PF-06438179 (N=323) | Period 1: Infliximab-EU Remicade (INX) (N=326) | Period 2: PF-06438179/PF-06438179 (N=280) | Period 2: INX/INX (N=143) | Period 2: INX/PF-06438179 (N=143) | Period 3: PF-06438179/PF-06438179/PF-06438179 (N=253) | Period 3: INX/INX/PF-06438179 (N=126) | Period 3: INX/PF-06438179/PF-06438179 (N=126)
Infusion related reaction (Injury, poisoning and procedural complications) | 19 | 21 | 8 | 11 | 6 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 19 | 15 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.